CLINICAL TRIAL: NCT04199299
Title: The Use of Sensors to Improve Communication for Persons With Intellectual Disability Who Cannot Communicate Unequivocally
Brief Title: Sensors for Communication for Persons Who Cannot Communicate Unequivocally
Status: Recruiting | Type: Observational
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Bjørnar Hassel, Professor, Senior consultant, University of Oslo
Other Study IDs: Understand me!
Record Dates: First submitted 2019-04-25; First posted 2019-12-13 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Intellectual Disability; Autism; Cerebral Palsy
MeSH Terms: conditions — Intellectual Disability; Autistic Disorder; Cerebral Palsy | interventions — Heart Rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons who cannot communicate unequivocally: Persons with intellectual disability, childhood autism, and/or cerebral palsy who cannot communicate unequivocally and therefore cannot communicate their needs and wishes, e.g. whether they are uncomfortable, in pain, scared, angry, happy, pleased.
  Interventions: Device: Heart rate and respiration rate sensors

INTERVENTIONS:
Device: Heart rate and respiration rate sensors — The use of sensors to monitor physiological variables (e.g. heart rate, sleep). The design is a before-and-after comparison with respect to whether the use of sensors has changed the caregivers' practice and their (perceived) understanding of the participant. The frequency of participants' self harm or aggressive behavior after as compared to before the introduction of pulse- and respiration monitors will also be charted.

SUMMARY:
Some persons with intellectual disability or comprehensive cerebral palsy cannot communicate unequivocally how they are, how they react to situations and people, whether they are in pain or experience discomfort, anger or fear. Their modes of communication (sounds, grimacing etc) may be unintelligible or ambiguous to their caregivers.

With the use of heart and/or respiration monitors the investigators aim to give these persons a means to communicate their immediate reactions or responses. The respiration monitor is meant to register sleep at night, so that the participants can communicate whether they have slept well or not the previous night.

DETAILED DESCRIPTION:
Heart rate (HR) is considered to reflect a persons autonomic response to situations, whether external (what happens around us) or internal (pain or pleasure, joy or fear). Some persons with severe intellectual disability or comprehensive cerebral palsy or childhood autism cannot communicate unequivocally, either because they lack the cognitive prerequisites and language or because they lack control over their muscles used for speech.

The investigators believe that these persons, through their heart rate, as registered with a commercially available chest belt or wrist watch, may communicate something about their well being and their reactions, preferences, aversions and fears.

Many persons with intellectual disability, comprehensive cerebral palsy or childhood autism (the participants in this study) have sleep problems, but these may go unnoticed. Participants often have a fixed schedule for the day, and this is carried out irrespective of the shape they are in, e.g. irrespective of how well they have slept the night before. The challenges may then be too much for a sleep-deprived person, and frustration and even self harm and aggressive behavior may be the result. With the use of a respiration monitor that assesses sleep from the person's breathing pattern, the person in question may be able to communicate to her/his caregivers how the previous night's sleep was.

Information about heart rate and sleep may contribute to better care and health services for persons who are unable to communicate unequivocally because of intellectual disability, autism and/or cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* intellectual disability with or without autism and/or cerebral palsy that render the participant unable to communicate his/her needs and reactions unequivocally.

Exclusion Criteria:

* allergic skin reaction to chest strap

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants are persons with intellectual disability (ID) and/or cerebral palsy (CP) that render the participant unable to communicate unequivocally. Participants with ID will typically have severe (IQ score 20-35) or profound (IQ score <20) ID. However, some may have moderate ID (IQ score 35-50) combined with autism of a degree that renders them unable to communicate unequivocally.
  Participants with CP typically have a severe variant that implies impaired control over muscles involved in communication (speech, gaze direction, gesticulation, pointing, mimic/grimacing), rendering them unable to communicate unequivocally. However, some participants with CP may also have ID, which contributes to the communication difficulties.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Caregivers' practice detailed in structured interview | 10 years
  Does the practice of the care for persons who cannot communicate unequivocally change after introduction of pulse- and respiration sensors? These questions are addressed in a structured interview with caregivers prior to and 2 months after the introduction of pulse- and respiration sensors.

SECONDARY OUTCOMES:
Caregivers' understanding of the user detailed in structured interview | 10 years
  Does introduction of pulse- and respiration sensors to allow participants to communicate pain, anxiety, sleeplessness etc., change caregivers' understanding of the participants' situation, needs and personality? These questions are addressed in a structured interview with caregivers prior to and 2 months after the introduction of pulse- and respiration sensors.

OTHER OUTCOMES:
Frequency of self harm or aggressive behavior measured by daily registration | 10 years
  Self harm and aggressive behavior are registered daily in the participants' dwellings, offering a means of comparing the frequency of such behavior before and after the introduction of pulse - and respiration sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørnar Hassel, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kildal ESM, Quintana DS, Szabo A, Tronstad C, Andreassen O, Naerland T, Hassel B. Heart rate monitoring to detect acute pain in non-verbal patients: a study protocol for a randomized controlled clinical trial. BMC Psychiatry. 2023 Apr 14;23(1):252. doi: 10.1186/s12888-023-04757-1. PMID 37060049
- [Background] Kildal E, Stadskleiv K, Boysen ES, Oderud T, Dahl IL, Seeberg TM, Guldal S, Strisland F, Morland C, Hassel B. Increased heart rate functions as a signal of acute distress in non-communicating persons with intellectual disability. Sci Rep. 2021 Mar 19;11(1):6479. doi: 10.1038/s41598-021-86023-6. PMID 33742078